CLINICAL TRIAL: NCT00541125
Title: Phase II, Multicenter Study Evaluating G-CSF as Primary Prophylaxis for Neutropenia Associated With First-line Chemotherapy Regimen FOLFIRI and Bevacizumab in Patients With Metastatic Colorectal Cancer Who Are Homozygous for UGT1A1*28 Polymorphism, the Promoter of the Gene Encoding for the Enzyme UGT1A1
Brief Title: G-CSF in Preventing Neutropenia During First-Line Treatment With Chemotherapy and Bevacizumab in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000564089; FFCD-0604; EU-20757; EUDRACT-2007-001772-37
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2016-05

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Filgrastim; Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRI-bévacizumab avec G-CSF en prophylaxie primaire (Other): FOLFIRI-bévacizumab avec G-CSF en prophylaxie primaire
  Interventions: Biological: bevacizumab; Biological: filgrastim; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Biological: bevacizumab
Biological: filgrastim
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: G-CSF may prevent or control neutropenia caused by first-line therapy in patients with metastatic colorectal cancer.

PURPOSE: This phase II trial is studying how well G-CSF works in preventing neutropenia during first-line treatment with chemotherapy and bevacizumab in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if primary prophylaxis comprising filgrastim (G-CSF) makes it possible to obtain neutropenia lower than grade 4 or a 30% decrease in fever in patients with metastatic colorectal cancer receiving first-line FOLFIRI and bevacizumab and who are homozygous for allele UGT1A1*28 (genotype 7/7), a promoter of the gene coding for enzyme UGT1A1.

Secondary

* Evaluate the objective response rate at 6 months of treatment with FOLFIRI and bevacizumab according to RECIST criteria.
* Evaluate the toxicity (excluding neutropenia) of FOLFIRI and bevacizumab according to NCI-CTC v. 2.0.
* Determine progression-free and overall survival.
* Determine the time to treatment failure.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes, irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1. Patients also receive filgrastim (G-CSF) subcutaneously on days 5-11. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 2-3 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Metastatic disease
  * Not surgically curable
* Homozygous for allele UGT1A1*28, the promoter of the gene coding for UGT1A1 (genotype 7/7)
* Measurable and/or evaluable disease

Exclusion criteria:

* Original tumor not removed
* CNS metastases
* Secondary localized cerebral tumors

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine > 1.5 mg/dL
* Total bilirubin ≤ 1.5 times normal
* Alkaline phosphatase ≤ 2.5 times normal (5 times normal if liver involvement)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients of must use effective contraception

Exclusion criteria:

* Progressive gastroduodenal ulcer, prior hemorrhagic ulcer, or perforation in the past 6 months
* Enteropathy or chronic diarrhea
* Chronic inflammatory intestinal disease
* Intestinal obstruction
* Active cardiac disease including any of the following:

  * Uncontrolled hypertension
  * Myocardial infarction in the past 12 months
  * Serious angina
  * NYHA class II-IV congestive heart failure
  * Severe arrhythmia (even if treated)
  * Peripheral vascular disease ≥ grade 2
* Unhealed wound, ulcer, or severe bone fracture
* Bleeding disorder or coagulopathy
* Severe uncontrolled infection or medical condition
* Proteinuria > 500 mg/24 hours
* Other malignancy within the past 5 years except basal cell skin cancer or curatively treated carcinoma in situ of the cervix
* Known dihydropyrimidine dehydrogenase deficiency
* Severe traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* At least 2 weeks since prior radiotherapy

Exclusion criteria:

* Prior chemotherapy for metastatic disease except adjuvant chemotherapy completed > 6 months ago
* Prior irinotecan hydrochloride or bevacizumab
* Major surgery or biopsy within the past 4 weeks
* Major surgery planned
* Puncture in the past week
* Chronic aspirin (> 325 mg/day) or NSAIDs
* Concurrent antifungal azoles (e.g., ketoconazole, fluconazole, itraconazole)
* Concurrent phenytoin (as in yellow fever vaccine)
* Concurrent Hypericum perforatum (St. John's wort)
* Oral or parenteral coagulant in the past 10 days and during study therapy

  * Warfarin allowed provided INR < 1.5

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of neutropenia grade 4 or fever | 2013
Toxicities by NCI-CTC v. 2.0 | 2013

SECONDARY OUTCOMES:
Objective response at 6 months by RECIST | 2013
Tolerance (except neutropenia) by NCI-CTC v. 2.0 | 2013
Progression-free survival | 2013
Overall survival | 2013
Time to treatment failure | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lecomte, MD, Study Chair — CHRU de Tours - Hopital Trousseau